CLINICAL TRIAL: NCT05115916
Title: Effect of Patient Portal Messaging Before Mailing Fecal Immunochemical Testing Kit on Colorectal Cancer Screening Rates: A Randomized Quality Improvement Trial
Brief Title: Effect of Patient Portal Messaging Before Mailing Fecal Immunochemical Testing Kit on Colorectal Cancer Screening Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: UCLA Vatche and Tamar Manoukian Division of Digestive Diseases (Unknown)
Responsible Party: Principal Investigator, Daniel M. Croymans, MD, MBA, MS, Medical Director, DOM Quality, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FITPrimer
Record Dates: First submitted 2021-10-28; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Cancer Screening
Keywords: Colorectal Cancer Screening; Colon Cancer; Nudge; Behavior and Behavior Mechanisms; Behavioral Economics; Health Screening
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Behavior

STUDY DESIGN:
Intervention Model Description: 3880 patients 51-75 years old, within the UCLA Health Managed Care group overdue for average risk CRC screening without prior history of documented FIT or colonoscopy will be randomized into 2 groups, in a 1:1 ratio. The 2 groups represent standard of care, and then the MyChart Message group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): This group will receive standard FIT mailer protocol (includes mailed FIT kit plus standardized messaging via EHR portal)
- MyChart Message (Experimental): This group will receive a message via EHR portal informing them about the incoming FIT Kit
  Interventions: Behavioral: MyChart Priming Message

INTERVENTIONS:
Behavioral: MyChart Priming Message — In addition to the standard FIT mailer protocol, we will send randomized participants a message via their personal health portal. Patients receive the primer approximately 1-2 weeks prior to arrival of the FIT kit, which informed patients about the incoming FIT Kit and instructed patients to complete and return the kit promptly.
  Arms: MyChart Message

SUMMARY:
Behavioral economics principles have increasingly been shown to improve health outcomes in the United States. They offer the ability to implement simple, low-cost and effective interventions to address key health issues without sacrificing the autonomy of patients. Colorectal cancer (CRC) screening is a key area where behavioral economics principles can help improve health outcomes. Despite being the second leading cause of cancer related death, the rate of CRC screening remains well below national targets. Interventions to address these issues, and improve screening rates at our institution have including implementing a Mailed FIT outreach program, and adding an informational letter that utilizes behavioral economic principles. To further improve our screening rates, this project builds upon our previous efforts to include a randomized electronic message primer via patients electronic patient portal, to help alert them of incoming FIT Kit and complete screening. This study will contribute to the growing literature of behavioral economics in medicine, while addressing an important health issue.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of death from cancers affecting both men and women in the United States. One in 17 Americans will suffer from CRC during his/her lifetime. Early detection by screening has been shown to reduce CRC mortality. Despite screening recommendations, the U.S. screening rate remains well below the national benchmark of 80% as established by the National Colorectal Cancer Roundtable. The U.S. Multi-Society Task Force (MSTF), however, does recommended FIT and colonoscopy as first line screening modalities for CRC in 2017. To help address the issue of suboptimal CRC screening, the investigators implemented an intervention utilizing the principles of behavioral economics to improve screening rates. Studies in behavioral economics and psychology indicate that how information or choice is framed impacts behavior in predictable ways, which has applications in health and medicine, including the design of CRC screening strategies. This project builds upon our institutions continued quality improvement efforts utilizing behavioral economics principles to improve CRC screening, through improving the choice architecture, framing and salience of information to incentivize routine screening.

For this project the investigators will leverage our electronic health records (EHR) patient portals to improve CRC screening. Specifically, the investigators developed an electronic primer within the EHR patient portal to alert patients due for CRC screening before arrival of a mailed FIT Kit. The investigators randomized implementation of the primer at the patient-level to determine whether the electronic primer improved CRC screening completion in patients enrolled in our mailed FIT program.

For our analysis, after summarizing our demographic data, the investigators plan to compare screening completion in the two study arms using an intention-to-treat analysis and t-tests. The investigators then plan a logistic regression and Cox proportional hazards model to compare time to screening utilization in the two study arms, controlling for age, sex, race, and ethnicity. Following this the investigators use Fisher's exact tests to compare completion of individual screening modalities in the two study arms. Lastly, the investigators plan a secondary, analysis to determine the impact of opening the portal message on screening utilization, using randomization arm as an instrumental variable. In this analysis the investigators compare the subset of patients in the intervention group that opened the portal primer message to the control group. P-values less than 0.05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Managed care patient, 51-75 years old
* Active primary care provider at UCLA seen within last 3 years

Exclusion Criteria:

* Inactive MyChart status or mailing address at time of enrollment
* Died within follow up period
* Any high-risk features including first degree family members with CRC, personal history of adenomas, history of inflammatory bowel disease, and any genetic GI cancer syndromes.
* Exclusion from March 2020 cohort if received FIT mailer within past 6 months

Ages: 51 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3880 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Overall Colorectal Cancer Screening Uptake | 6 months
  Rate of completion of CRC screening by any of the following: FIT, colonoscopy, CT colonography, sigmoidoscopy or FIT-DNA within study period.

SECONDARY OUTCOMES:
Time to screening | 6 months
  Time (months) to screening uptake
Colorectal cancer screening uptake by modality | 6 months
  Rate of completion of CRC screening by modality type
Effect of electronic primer message on CRC uptake among participants who opened | 6 months
  Rate of completion of CRC screening among individuals who received the MyChart electronic primer.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Westwood, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD for this investigation.

REFERENCES:
- [Derived] Goshgarian G, Sorourdi C, May FP, Vangala S, Meshkat S, Roh L, Han MA, Croymans DM. Effect of Patient Portal Messaging Before Mailing Fecal Immunochemical Test Kit on Colorectal Cancer Screening Rates: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2146863. doi: 10.1001/jamanetworkopen.2021.46863. PMID 35119462